CLINICAL TRIAL: NCT00614640
Title: A Phase I/II Study of the Safety, Tolerability, and Immunogenicity of a Topical Therapeutic DNA Dendritic Cell Vaccine (DermaVir Patch) in Children, Adolescents, and Young Adults With HIV-1 Infection on Highly Active Antiretroviral Therapy (HAART)
Brief Title: Safety and Tolerability of a Therapeutic DNA Dendritic Cell Vaccine in HIV-Infected Children, Adolescents, and Young Adults
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1049; 10165 (Registry Identifier: DAIDS ES Registry Number); IMPAACT P1049
Record Dates: First submitted 2008-02-11; First posted 2008-02-13 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HAART; Therapeutic vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): One 0.8 ml vaccine-containing patch and 1 placebo patch placed on upper back or upper thigh for 24 hours on Days 0, 42, and 84
  Interventions: Biological: DermaVir patch; Biological: Placebo patch
- 2 (Experimental): Four 0.8 ml vaccine-containing patches placed on upper back or upper thigh for 24 hours on Days 0, 42, and 84
  Interventions: Biological: DermaVir patch
- 3 (Experimental): Four 0.8 ml vaccine-containing patches placed on upper back or upper thigh for 24 hours on Days 0, 7, 42, 49, 84, and 91
  Interventions: Biological: DermaVir patch

INTERVENTIONS:
Biological: DermaVir patch — DNA Vaccine
  Other Names: LC002
Biological: Placebo patch — 10% dextrose (D-glucose) solution
  Other Names: LC002 placebo
  Arms: 1

SUMMARY:
The therapeutic DNA vaccine, DermaVir, represents an immunization strategy that targets lymph node dendritic cells. Because of the high percentage of naive CD4 cells in children and adolescents, the potential for effective new HIV-specific CD4 cell responses may be more achievable in children than in adults. The primary purpose of this study is to evaluate the safety and tolerability of DermaVir in children and young adults.

DETAILED DESCRIPTION:
The introduction of highly active antiretroviral therapy (HAART) for children and adolescents has resulted in improved control of viral replication for prolonged periods of time and a significant reduction in morbidity. However, when compared to the responses seen in adults, children have overall inferior virologic responses. The therapeutic vaccine, DermaVir, represents an immunization strategy that targets lymph node dendritic cells. Because of the high percentage of naive CD4 cells in children and adolescents, the potential for effective new HIV-specific CD4 cell responses may be more achievable in children than in adults. The primary purpose of this study is to evaluate the safety and tolerability of DermaVir in children and young adults.

This study will last up to 61 weeks (up to 13 weeks of treatment with an additional 48 weeks for follow-up). Participants will be randomly stratified according to age and dosage. Group 1 will consist of 8 adolescents and young adults (between ages 13 and 23) and 8 children (between ages 6 and 12). Group 1 participants will have one 0.8 ml DermaVir patch and one control patch applied on Days 0, 42, and 84. Group 2 will consist of 4 adolescents and young adults and 4 children. Group 2 participants will have four 0.8 ml DermaVir patches applied on Days 0, 42, and 84. Group 3 will consist of 4 adolescents and young adults and 4 children. Group 3 participants will have four 0.8 ml DermaVir patches applied on Days 0, 7, 42, 49, 84, and 91.

There will be 14 study visits for each participant. They will occur at screening and Days 0, 7, 21, 42, 49, 63, 84, 91, 105, 126, 168, 259, and 427. Screening will occur up to 30 days before the first vaccination (Day 0). Medical history and physical exam will occur at all visits. Blood and urine collection and an adherence assessment will occur at most visits. A urine pregnancy test will occur for females at most visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Receiving HAART consisting of drugs from at least 2 different classes for at least 12 months prior to study entry
* CD4 count of 350 cells/mm3 or greater
* Viral load less than 400 copies/ml for at least 12 months prior to screening
* If female, agree to avoid pregnancy and use two methods of contraception. More information on this criterion can be found in the protocol.
* If male, agree to avoid attempting to impregnate a female and not participate in sperm donation programs. Male participants must agree to use a condom during sexual activity from the date of receipt of the first study vaccination until 6 months after receipt of the last study vaccination.

Exclusion Criteria:

* Failing antiretroviral regimen
* Skin diseases, including active atopic dermatitis, active or history of psoriasis, active urticaria, known hypersensitivity to adhesive tape, history of keloid, and active or history of vitiligo
* Tattoos or changes in pigment at selected skin vaccination sites
* Hair or tattoo removal in close proximity to vaccine site on skin
* Acute or chronic illness. More information on this criterion can be found in the protocol.
* Chronic autoimmune disease, clinically significant bleeding disorder, or insulin dependent diabetes mellitus
* Clinical toxicity (Grade 2 or greater) at screening
* Prior treatment with any HIV vaccine
* Treatment with any HIV immune modulating agents or chemotherapy for malignancy within 12 months of study entry
* Vaccinations within 28 days of study entry
* Participation in an investigational new drug protocol within 60 days prior to screening
* Systemic steroid therapy within 28 days of study entry
* Abnormal laboratory values. More information on this criterion can be found in the protocol.
* Excessive exposure to the sun
* Breastfeeding or pregnant

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Suspected adverse drug reaction (SADR) attributable to vaccine, excluding reaction to patch adhesive | Throughout study
Toxicity attributable to the adhesive on patch and not to the vaccine product | Throughout study
Decrease in CD4 count by 1/3 of baseline in 2 separate measurements at least 1 month apart | Throughout study
Viral load greater than 1000 copies/ml on 2 separate measurements at least 2 weeks apart | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Hans M.L. Spiegel, MD, Study Chair — George Washington University School of Medicine; Willaim Borkowsky, MD, Study Chair — NYU Langone Health; Ram Yogev, MD, Study Chair — CMRC Children's Memorial Hospital; Elizabeth McFarland, MD, Study Chair — University of Colorado Health Sciences Ctr.

REFERENCES:
- [Background] Calarota SA, Weiner DB, Lori F, Lisziewicz J. Induction of HIV-specific memory T-cell responses by topical DermaVir vaccine. Vaccine. 2007 Apr 20;25(16):3070-4. doi: 10.1016/j.vaccine.2007.01.024. Epub 2007 Jan 22. PMID 17292518
- [Background] Lisziewicz J, Calarota SA, Lori F. The potential of topical DNA vaccines adjuvanted by cytokines. Expert Opin Biol Ther. 2007 Oct;7(10):1563-74. doi: 10.1517/14712598.7.10.1563. PMID 17916048
- [Background] Lori F, Weiner DB, Calarota SA, Kelly LM, Lisziewicz J. Cytokine-adjuvanted HIV-DNA vaccination strategies. Springer Semin Immunopathol. 2006 Nov;28(3):231-8. doi: 10.1007/s00281-006-0047-y. Epub 2006 Oct 20. PMID 17053912